CLINICAL TRIAL: NCT02318186
Title: Multi-center, Open-label Pharmacokinetic Study of Subcutaneously and Intravenously Administered Treprostinil in Children With Pulmonary Arterial Hypertension (PAH)
Brief Title: Pharmacokinetic Study of Sub-q and IV Treprostinil in Kids With Pulmonary Arterial Hypertension (PAH)
Acronym: PKRemodulin
Status: Completed | Type: Observational
Sponsor: Jeffrey A. Feinstein (Other)
Collaborators: United Therapeutics (Industry); Seattle Children's Hospital (Other); University of Colorado, Denver (Other); Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor-Investigator, Jeffrey A. Feinstein, Director, Vera Moulton Wall Center for Pulmonary Vascular Disease, Stanford University
Organization: Stanford University (Other)
Other Study IDs: UT PK Treprostinil
Record Dates: First submitted 2014-01-09; First posted 2014-12-17 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pharmacokinetic analysis; remodulin; trepostinil; pulmonary arterial hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 2 mL blood sample in K3-EDTA tube and immediately place on ice; Place plasma into 2 aliquots; Freeze at -20 degrees or lower. Store until batch is complete; Batch ship all samples on dry ice to pharmacokinetic analytical laboratory
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- 0 months - 1 year
- 11-16 years
- 7-11 years
- 4-6 years
- 1-3 years

SUMMARY:
Abstract

This is a multi-center, open-label pharmacokinetic (PK) study examining the relationship between the steady-state plasma concentration and dose of treprostinil delivered intravenously or subcutaneously in children with pulmonary arterial hypertension (PAH). Subjects will be divided into 5 cohorts by age. A blood sample will be obtained from each subject at steady state. Additional blood samples will be obtained from a small subset of subjects with a 15% increase or with at least a 15ng/kg/min increase in dose from steady state. Samples will be sent to a pharmacokinetic laboratory for analysis. Linear regression analysis will be used to determine the relationship between the steady state plasma concentration and drug dose. A power model will be used to assess dose proportionality.

DETAILED DESCRIPTION:
Background Information and Rationale

Treprostinil has not been adequately studied to determine its safety and efficacy in children ≤ 16 years old. However, the drug's use and tolerance in children with PAH has been demonstrated in studies with small sample sizes.

Although the pharmacokinetic relationship of treprostinil has been established in adult patients with PAH, the relationship between the steady-state plasma concentration and dose for children requires further investigation because of physiologic differences, such as the maturity of enzyme systems and drug clearance mechanisms, between children and adults. The subjects in this study will be divided into cohorts by age to address the physiologic changes that occur throughout childhood.

Currently, no data exists demonstrating the relationship between the steady-state plasma concentration and dose for children treated with intravenously or subcutaneously delivered treprostinil. Understanding the pharmacokinetics of treprostinil among different age cohorts in children will provide the data to make an informed recommendation for dosing based on age (and possibly weight).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be on continuous intravenous or subcutaneous treprostinil for the treatment of pulmonary arterial hypertension, defined as mean pulmonary artery pressure >25mmHg at rest with a PVRi > 3 Wood units.
2. Patients must be between the ages of 0 to 16 years at the time of study enrollment.
3. Written informed consent and assent, when applicable, must be completed.

Exclusion Criteria:

1. Patients with severe liver or renal diseases.
2. Female patients who may be pregnant or breastfeeding
3. Written informed consent and assent not completed due to patient and/or parent or legal guardian unwilling to participate.
4. Patients on concomitant use of a CYP2C inhibitor or inducer.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Target enrollment for this study is a total of 50 pediatric patients among all participating sites with a goal of 65 total blood samples. Cohorts will be: 0-12 months; 1-3 years; 4-6 years; 7-11 years; 11-16 years. Each cohort will have 10 patients with 5 patients on a dose ≤ 50ng/kg/min and 5 patients on a dose ≥51-120ng/kg/min.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2013-10; Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
To determine the relationship between steady-state plasma concentration and dose of treprostinil within each age cohort and among age cohorts. | at least 48 hours after most-recent titration
  A blood sample will be obtained from each subject at steady state. Additional blood samples will be obtained from a small subset of subjects with a 15% increase or with at least a 15ng/kg/min increase in dose from steady state.

SECONDARY OUTCOMES:
To correlate PK level of treprostinil with the presence or absence of side effects | At time of blood draw
  A survey of side effects (GI, neurological, cardiac, respiratory, skin) will be administered at time of blood draw.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Feinstein, MD, MPH, Principal Investigator — Stanford University
Locations (1):
- Lucille Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Publication

REFERENCES:
- [Background] Ivy DD, Claussen L, Doran A. Transition of stable pediatric patients with pulmonary arterial hypertension from intravenous epoprostenol to intravenous treprostinil. Am J Cardiol. 2007 Mar 1;99(5):696-8. doi: 10.1016/j.amjcard.2006.09.119. Epub 2007 Jan 10. PMID 17317374
- [Background] Levy M, Celermajer DS, Bourges-Petit E, Del Cerro MJ, Bajolle F, Bonnet D. Add-on therapy with subcutaneous treprostinil for refractory pediatric pulmonary hypertension. J Pediatr. 2011 Apr;158(4):584-8. doi: 10.1016/j.jpeds.2010.09.025. Epub 2010 Oct 30. PMID 21035821
- [Background] McSwain CS, Benza R, Shapiro S, Hill N, Schilz R, Elliott CG, Zwicke DL, Oudiz RJ, Staszewski JP, Arneson CP, Wade M, Zaccardelli D, McLaughlin V. Dose proportionality of treprostinil sodium administered by continuous subcutaneous and intravenous infusion. J Clin Pharmacol. 2008 Jan;48(1):19-25. doi: 10.1177/0091270007309708. PMID 18094217